CLINICAL TRIAL: NCT01326026
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec Once Daily in Insulin naïve Subjects With Type 2 Diabetes Mellitus When Titrated Using Two Different Titration Algorithms (BEGIN™: ONCE SIMPLE USE)
Brief Title: Comparing the Efficacy and Safety of NN1250 Once Daily When Titrated Using 2 Different Algorithms in Insulin naïve Subjects With Type 2 Diabetes Mellitus
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3846; U1111-1117-0616 (Other: WHO); 2010-022337-29 (EudraCT Number)
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg Simple (Experimental)
  Interventions: Drug: insulin degludec
- IDeg Step wise (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily. Dose individually adjusted.
  Arms: IDeg Simple
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily. Dose individually adjusted in a stepwise manner.
  Arms: IDeg Step wise

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to compare the efficacy and safety of NN1250 (insulin degludec (IDeg)) once daily in insulin naïve subjects with type 2 diabetes mellitus when titrated using two different self-titration algorithms (dose individually adjusted) in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 24 weeks prior to randomisation (Visit 2)
* Current treatment: metformin monotherapy or metformin in any combination with 1 or 2 other OADs including an insulin secretagogue (sulfonylurea or glinide), dipeptidyl peptidase IV (DPP-IV) inhibitors, alpha-glucosidase inhibitors, thiazolidinediones (TZDs) all with unchanged dosing for at least 12 weeks prior to randomisation (Visit 2)-metformin: alone or in combination (including fixed combination) must be at least 1000 mg daily
* HbA1c 7.0-10.0% (both inclusive) by central laboratory analysis
* BMI (Body Mass Index) no higher than 45.0 kg/m^2

Exclusion Criteria:

* Treatment with glucagon-like peptide 1 (GLP-1) receptor agonist within the last 12 weeks prior to Visit 2
* Suffer from a life threatening disease (e.g. cancer)
* Females of childbearing potential who are pregnant (as determined by central laboratory beta-human chorionic gonadotropin (beta-hCG), breast feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive methods as required by law or practise [for Germany, adequate contraceptive methods are: implants, injectables, combined oral contraceptives, hormonal IUD, sexual abstinence or vasectomised partner])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (43):
- United States (27):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, National City, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Killeen, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- Germany (6):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Völklingen
- Spain (6):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Antequera
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón

REFERENCES:
- [Result] Philis-Tsimikas A, Brod M, Niemeyer M, Ocampo Francisco AM, Rothman J. Insulin degludec once-daily in type 2 diabetes: simple or step-wise titration (BEGIN: once simple use). Adv Ther. 2013 Jun;30(6):607-22. doi: 10.1007/s12325-013-0036-1. Epub 2013 Jun 29. PMID 23812875
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 43 sites in 4 countries: Finland (5), Germany (6), Spain (6) and United States of America (26).
Pre-assignment Details: Subjects continued on metformin treatment at the pre-randomisation dose level and dosing frequency.
Groups:
- IDeg Simple: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (approximately 8-40 hours intervals between doses) with pre-trial metformin according to simple titration algorithm: self-titration was performed once weekly based upon a single pre-breakfast self measured plasma glucose (SMPG) value measured on the day of insulin titration.
- IDeg Step Wise: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (approximately 8-40 hours intervals between doses) with pre-trial metformin according to step wise titration algorithm: self-titration was performed once weekly based on the lowest value of three pre-breakfast SMPG values measured on three consecutive days, the two days prior to and on the day of insulin titration.
Period: Overall Study
Arm/Group | IDeg Simple | IDeg Step Wise
Started | 111 | 111
Exposed | 110 (One subject withdrew before exposure to trial drug) | 111
Completed | 99 | 98
Not Completed | 12 | 13
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal Criteria | 5 | 7
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg Simple | IDeg Step Wise | Total
Number analyzed (Participants) | 111 | 111 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.5) | 58.5 (11.1) | 58.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 79
  Male | 68 | 75 | 143
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.1 (0.9) | 8.2 (0.9) | 8.1 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.3 (2.6) | 9.4 (2.8) | 9.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg Simple | IDeg Step Wise
Number analyzed (Participants) | 111 | 111
percentage of glycosylated haemoglobin | -1.09 (1.05) | -0.93 (0.97)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). For 7 subjects baseline values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg Simple | IDeg Step Wise
Number analyzed (Participants) | 108 | 107
mmol/L | -3.27 (3.56) | -2.68 (3.50)

3. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDeg Simple | IDeg Step Wise
Number analyzed (Participants) | 110 | 111
Events/100 years of patient exposure
  Adverse events (AEs) | 346 | 379
  Serious AEs | 15 | 15
  Severe AEs | 15 | 10
  Moderate AEs | 69 | 79
  Mild AEs | 262 | 291
  Fatal AEs | 0 | 2

4. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Observed rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg Simple | IDeg Step Wise
Number analyzed (Participants) | 110 | 111
Episodes/100 years of patient exposure | 160 | 117

5. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Observed rate of nocturnal confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg Simple | IDeg Step Wise
Number analyzed (Participants) | 110 | 111
Episodes/100 years of patient exposure | 21 | 10

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: The safety analysis set included all subjects who received at least one dose of the investigational product.
Arm/Group | IDeg Simple | IDeg Step Wise
Serious Adverse Events (participants affected / at risk) | 5/110 | 7/111
Other Adverse Events (participants affected / at risk) | 17/110 | 14/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg Simple (N=110) | IDeg Step Wise (N=111)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg Simple (N=110) | IDeg Step Wise (N=111)
Nasopharyngitis (Infections and infestations) | 10 (10) | 7 (8)
Headache (Nervous system disorders) | 8 (8) | 8 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.